CLINICAL TRIAL: NCT02096536
Title: Exploring Vancomycin Disposition in Neonates: Paired Analysis of Vancomycin Concentrations Using Immunoassay and Liquid-chromatography-tandem Mass Spectrometry. Determination of Vancomycin Protein Binding and Its Covariates in Neonates
Brief Title: Exploring Vancomycin Disposition in Neonates
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S56376
Record Dates: First submitted 2014-03-17; First posted 2014-03-26 (Estimated); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Neonatal Infection
Keywords: Neonate; Vancomycin; LC/MS-MS; protein binding
MeSH Terms: interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vancomycin (Other): All included patients receive vancomycin for medical reasons. Decision for start of therapy is made by the treating physician.
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — vancomycin administration based on decision of treating physician
  Other Names: Vancomycine Actavis

SUMMARY:
Vancomycin is already used for decades in neonates. However, there are remaining questions concerning vancomycin disposition in this population. The purpose of this study is first of all to perform a paired analysis of serum vancomycin concentrations using an immunoassay versus a reference liquid chromatography-tandem mass spectrometry method. Secondly, we aim to determine vancomycin protein binding and its covariates in neonates.

DETAILED DESCRIPTION:
Exploration of vancomycin disposition in neonates:

Objective 1: Paired analysis of (total) serum vancomycin concentrations in neonates using the currently available immunoassay (Cobas c702) versus a reference liquid chromatography-tandem mass spectrometry method (LC-MS/MS).

Objective 2: The determination of vancomycin protein binding and its covariates in neonates.

ELIGIBILITY:
Inclusion Criteria:

* Neonates, admitted to the Neonatal Intensive Care Unit to whom vancomycin is administered for medical reasons, can be included in the study after informed consent of the parents.

Exclusion Criteria:

* No vancomycin therapy
* No signed informed consent available

Ages: 1 Day to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2014-04; Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Differences in vancomycin exposure | 1 year
  Paired vancomycin concentrations in 60 neonates using an immunoassay versus LC/MS-MS method.
  Total versus unbound vancomycin concentrations in 60 neonates.

SECONDARY OUTCOMES:
Impact of freezing and thawing on vancomycin measurement | 1 year
  Comparisson of the same analytical technique (immunoassay) in fresh (routine clinical care) versus stored samples .

CONTACTS AND LOCATIONS:
Overall Officials: Anne Smits, MD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium